CLINICAL TRIAL: NCT06708975
Title: Effect of Transdermal Insulin Therapy by Ultrasonographic in Wound Healing of Chronic Diabetic Patients
Brief Title: Effect of Insulin Therapy by Ultrasonography in Wound Healing of Chronic Diabetic Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Radwa Fayek Hammam, Lecturer at Basic Science Department, Faculty of Physical Therapy Modern University for Technology and Information, MTI University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P.T.REC/012/005342
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellites, Insulin Phonophoresis
MeSH Terms: conditions — Diabetes Mellitus | interventions — Bandages

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): subjects will receive Phonophoresis Insulin Therapy, hyperpolarized light therapy and Standard wound cleaning and dressing.
  Interventions: Other: Insulin therapy phonophoresis; Other: Hyperpolarized light therapy and Standard wound cleaning and dressing.
- Group B (Sham Comparator): subjects will receive hyperpolarized light therapy and Standard wound cleaning and dressing
  Interventions: Other: Hyperpolarized light therapy and Standard wound cleaning and dressing.

INTERVENTIONS:
Other: Insulin therapy phonophoresis — Insulin therapy phonophoresis is the use of ultrasound to deliver drugs through patients skin, Insulin therapy will be used to determine its effect on wound healing in patients with chronic diabetes mellites because in addition to its systemic impact, numerous reports suggest that applying insulin topically causes localized effects. Many trials and case reports have been released reporting positive effects of topical insulin for many diseases such as dermatological compromises, ophthalmological diseases and others
  Arms: Group A
Other: Hyperpolarized light therapy and Standard wound cleaning and dressing. — Hyperpolarized light therapy safely accelerates wound healing by stimulating blood circulation, reducing inflammation and relieving muscle spasms.

SUMMARY:
The main aim of the study is to determine the effect of transdermal application of insulin therapy by phonophoresis in wound healing in diabetic patients the main question of the study: is insulin phonophoresis is effective in accelerating healing in patients with diabetes mellites? 40 patients will be randomly assigned to two groups group A will receive insulin phonophoresis plus hyper polarized laser therapy and standard wound cleaning and dressing three times weekly over four weeks.

Group B will receive hyper polarized laser therapy and standard wound cleaning and dressing three times weekly over four weeks.

DETAILED DESCRIPTION:
DIMST scale ( as an acronym from the initial domains of depth, maceration, inflammation/infection, size, tissue type of the wound bed, type of wound edge, and tunneling/undermining) will be used for assessment.

MANOVA will be used for statistical analysis between group comparison

ELIGIBILITY:
Inclusion Criteria:

* patients will be included if they are free from any pathological condition like limb infection, local or proximate malignancy, and anti-coagulated patients.

Exclusion Criteria:

patients will be excluded if they have any pathological condition like limb infection, local or proximate malignancy, and anti-coagulated patients.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
DMIST scale which is a valid and reliable scale for measuring depth, maceration, inflammation/infection, size, tissue type of the wound bed, type of wound edge, and tunneling/undermining. | before first session and at the end of the treatment program (four weeks)
  Zero will be the minimum score and 98 was the maximum, with a greater number denoting a more severe injury and a zero signaling full recovery

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: EFFECT OF TRANSDERMAL INSULIN DELIVERY BY LOW INTENSITY ULTRASOUND IN HEALING OF CHRONIC LOWER LIMB VENOUS ULCER — https://fizjoterapiapolska.pl/en/article/wplyw-przezskornego-podawania-insuliny-za-pomoca-ultradzwiekow-o-niskiej-intensywnosci-na-gojenie-przewleklego-owrzodzenia-zylnego-konczyn-dolnych/